CLINICAL TRIAL: NCT00638144
Title: Prevention of Graft Reinfection After Liver Transplantation for HCV Related End-stage Liver Disease . Study of Humoral Anti-HCV Response
Brief Title: Prevention of Graft Reinfection After Liver Transplantation With Anti HCV Monoclonal Antibodies Identified in Chronically Infected Patients or in Patients With Resolved Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4109
Record Dates: First submitted 2008-03-03; First posted 2008-03-18 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; liver transplantation; antibodies mediated neutralization; monoclonal antibodies
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with resolved infection
- 2: chronically infected patients

SUMMARY:
End stage HCV-related cirrhosis has become a major indication for liver transplantation (LT). Unfortunately, recurrence of HCV infection on the liver graft occurs in almost all patients following transplantation and causes a persistent infection that leads to chronic hepatitis and cirrhosis in a significant proportion of patients. To date there is no effective way to prevent HCV reinfection of the liver graft in the early phase after transplantation. . Early passive immunotherapy with neutralizing antibodies against HCV should be considered for preventing reinfection of liver transplanted patients associated with HCV. This approach is well established in the case of patients undergoing liver transplantation for chronic hepatitis B virus infection. Our purpose is to produce neutralizing monoclonal antibodies to prevent reinfection of the liver graft.

ELIGIBILITY:
Inclusion Criteria:

* Health insurance
* Resolved HCV infection ( HCV RNA negative since more then 6 months ) -HCV chronically infected ( RNA positive )
* Anti- HCV antibodies positive
* Volunteers and informed patients

Exclusion Criteria:

* Immunosuppression
* HBV or HIV infection
* Pregnancy
* Breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with resolved infection chronically infected patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michel DOFFOEL, MD, Principal Investigator — CHRU Strasbourg; Albert FARADJI, MD, Principal Investigator — CHRU Strasbourg; Philippe WOLF, MD, Principal Investigator — CHRU Strasbourg
Locations (3):
- France (3):
  - Service d'Hépato-Gastro-Entérologie - Hôpital Civil, Strasbourg
  - Service d'Hématologie et Oncologie - Hôpital de Hautepierre, Strasbourg
  - Service de Chirurgie Générale et Transplantation Multiorganes - Hôpital de Hautepierre, Strasbourg